CLINICAL TRIAL: NCT03776565
Title: Gastric Ultrasound Before Planned Caesarean Section or Operative Hysteroscopy : How Much Pregnancy Changes Surface of Antrum of the Stomach ? Comparative Observational Study
Brief Title: Comparison of Antrum Surface Between Women With Operative Hysteroscopy or Planned Caesarean Section
Acronym: ECHOCESAR
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2017029F
Record Dates: First submitted 2018-11-26; First posted 2018-12-14 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Pregnancy Related
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Operative hysteroscopy: women with an operative hysteroscopy planned
  Interventions: Other: Ultrasound
- Planned caesarean section: Pregnant women with a planned caesarean section
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Ultrasound — Ultrasound of antrum of stomach

SUMMARY:
Realization of a gastric ultrasound just before surgery, to measure the surface of antrum of stomach and compare if divergence sizes can be observed between women with a operative hysteroscopy and women with a planned caesarean section. To know if anaesthesia need to be adapted to the population.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40
* Membership of a national insurance scheme
* Written consent
* Physical status score or American Society of Anesthesiologists (ASA) score = 1 or 2
* Planned caesarean section or operative hysteroscopy

Exclusion Criteria:

* Not able to give her written consent (not speaking French), under legal protection
* Insulin-dependant diabetes
* Hiatus hernia
* History of gastro-oesophageal surgery
* Contraindication to right lateral decubitus
* Treatments with anti-acids before ultrasounds.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Women comming to hospital/sites for a planned caesarean section or operative hysteroscopy.
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
Measure of antral surface | Just before anesthesia and surgery
  Measure of gastric antrum surface by Ultrasound on operative hysteroscopy women and planned caesarean section women.

SECONDARY OUTCOMES:
Measure of Perlas score | Before surgery
  Perlas score (Grade 0, defined as an empty antrum in both the supine and the right lateral decubitus positions, indicates that the stomach is completely empty; grade 1, defined as visualisation of gastric fluid content in the right lateral position only, corresponds to low gastric fluid volume; grade 2, defined by visualisation of liquid contents in both supine and right lateral positions, suggests a high gastric fluid volume with increased risk for pulmonary aspiration) measure by Ultrasound on operative hysteroscopy women and planned caesarean section women.
Assessment of anxiety on gastric residue with a numeric scale | Before surgery
  Measure of anxiety with a numeric scale (0 = no anxiety, 10 = maximal anxiety)
Assessment of frequency of intraoperative inhalation | During surgery
  Comparison of proportion of inhalation between the two population
Incidence of fasting on gastric residue between the two populations | Before surgery
  Comparison of antral surface with fasting as covariable

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Mercier, MD PhD, Study Director — Hopital Beclere (APHP)
Locations (2):
- France (2):
  - Hopital Béclère (APHP), Clamart
  - Hopital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No